CLINICAL TRIAL: NCT02845349
Title: Vortioxetine for the Treatment of Major Depression and Neuropsychiatric Co-morbidities After Traumatic Brain Injury (TBI)
Brief Title: Vortioxetine for the Treatment of Major Depression and Co-morbidities After Traumatic Brain Injury (TBI)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding withdrawn.
Sponsor: Johns Hopkins University (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00105196
Record Dates: First submitted 2016-07-18; First posted 2016-07-27 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: TBI; Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug-Vortioxetine (Experimental): The treatment group will receive vortioxetine 10 mg per day, which will be increased to 20 mg or decreased to 5 mg, if deemed clinically necessary, at week 4 or 8.
  Interventions: Drug: Vortioxetine
- Placebo (Placebo Comparator): Matching placebo will be used.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vortioxetine — The study drug, vortioxetine received approval from the U.S. Food and Drug Administration (FDA) to treat adults with major depressive disorder. This study is being done to determine its effectiveness in a specialized population, i.e. those who have developed major depression after a traumatic brain injury. As patients who have sustained a TBI are medically fragile and sensitive to side-effects of medications, it is important to test the effectiveness and safety of vortioxetine in this population.
  Other Names: Trintellix
  Arms: Drug-Vortioxetine
Drug: Placebo — A placebo comparator will be used in one subset of patients.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Traumatic brain injury (TBI) is a major public health problem with an annual incidence of about 1.7 million per year. TBI is associated with various long-term morbidities. Among them, psychiatric disturbances are the major cause of chronic disability and poor quality of life. Major depression is the common psychiatric sequela post TBI with rates ranging from 13% at 1 year to 60% at 8 years after TBI. Major depression after TBI (henceforth referred to as TBI depression) is often associated with comorbid neuropsychiatric symptoms (NPS) such as anxiety, aggression, substance abuse and cognitive deficits that often makes treatment difficult. Despite increased rates of depression, there is no Food and Drug Administration (FDA) approved drug/s for its treatment.

The investigators propose to address these limitations by use of a novel serotonergic agent, vortioxetine, which has a multimodal mechanism of action through serotonin transporter (SERT) inhibition, 5-hydroxytryptamine (5-HT)3, 7, and 1D receptor antagonism, 1B receptor partial agonism, and 1A receptor agonism.

Overarching Goal: The overarching goal of the proposed pilot study is to determine the effectiveness and safety of vortioxetine for the treatment of post-TBI depression and co-morbid NPS.

Study Design: The study design will include a DBPCT of 30 TBI patients of all severities who meet the DSM 5 criteria for major depression. A total of 150 will be consented to allow for screen failures. Written informed consent will be obtained from these patients. Subjects will be followed for a total of 12 weeks. Subjects will be randomized to either the vortioxetine arm (N=15) or placebo arm (N=15). The treatment group will receive vortioxetine 10mg per day, which will be increased to 20 mg or decreased to 5 mg, if deemed clinically necessary, at week 4 or 8. Subjects will have a total of 4-5 visits: Baseline evaluation (1 or 2 visits) and follow-up visits at weeks 4, 8 and 12. Well-validated psychiatric instruments will be used to compare the effectiveness of vortioxetine versus placebo treatment at week 12 compared to baseline Relevance: This study has the potential to provide strong preliminary evidence for the use of vortioxetine as a safe and novel agent for treatment of TBI depression and its psychiatric co-morbidities. If found to be effective, results from this study can be used to design larger studies and also determine brain changes associated with its use via neuroimaging.

DETAILED DESCRIPTION:
In this study the investigators propose to recruit 30 outpatients with TBI of varying degrees of severity who also meet DSM 5 criteria for major depression. The investigators will screen as many potential subjects as possible to get a total of 30 participants who meet the study criteria and complete the study ( Total 30 study completers). Written informed consent will be obtained from all participants prior to collection of any data. Participants will be evaluated using well validated psychiatric instruments Participants will be recruited from several sources: (1) Brain Injury Clinic at Johns Hopkins Bayview Medical Center; (2) referral from other Hopkins outpatient clinics; (3) Brain injury support groups organized by the Brain Injury Association of Maryland, and (4) Advertisements placed in local newspapers and (5) Trial Facts - an online recruiting source. The study sites will be at the Geriatric & Neuropsychiatry clinics at Johns Hopkins Bayview Medical Center.

Overarching Goal: The overarching goal of the proposed pilot study is to determine the effectiveness and safety of vortioxetine for the treatment of post-TBI depression and co-morbid neuropsychiatric symptoms (NPS).

Study Design: The study design will include a Double Blinded Placebo Controlled Trial (DBPCT) of 30 TBI patients of all severities who meet the DSM 5 criteria for major depression. A total of 150 will be consented to allow for screen failures. Written informed consent will be obtained from these patients. Subjects will be followed for a total of 12 weeks. Subjects will be randomized to either the vortioxetine arm (N=15) or placebo arm (N=15). The treatment group will receive vortioxetine 10mg per day, which will be increased to 20 mg or decreased to 5 mg, if deemed clinically necessary, at week 4 or 8. Subjects will have a total of 4-5 visits: Baseline evaluation (1 or 2 visits) and follow-up visits at weeks 4, 8 and 12.

Well-validated psychiatric instruments will be used to compare the effectiveness of vortioxetine versus placebo treatment at week 12 compared to baseline for the treatment of major depression and its neuropsychiatric co-morbidities.

Relevance: This study has the potential to provide strong preliminary evidence for the use of vortioxetine as a safe and novel agent for treatment of TBI depression and its psychiatric co-morbidities. If found to be effective, results from this study can be used to design larger studies and also determine brain changes associated with its use via neuroimaging. Depression is common in other neurological disorders such as stroke, multiple sclerosis, Parkinson's disease, and dementia syndromes. Results from this study can shed light in the management of depression in other neurological disorders.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over
* Meet Department of Defense Criteria for TBI
* Meet DSM 5 criteria for major depression
* Score greater than 16 on the HAM D17
* Currently not on any psychotropics for treatment of depression

Exclusion Criteria:

* Subjects who are medically or psychiatrically unstable
* Pregnant women
* History of active substance abuse x 1 month
* Other neurological problems, or a diagnosis of schizophrenia, dementia, or bipolar disorder
* Prior treatment with vortioxetine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Reduction of depressive symptoms at 12 weeks as assessed by the Hamilton Depression Scale 17 items (HAMD-17) | at 12 weeks
Reduction of depressive symptoms at 12 weeks as assessed by the Clinical Global Impression Improvement (CGI-I) scale | at 12 weeks

SECONDARY OUTCOMES:
Comparison of rates and severity of side-effects and adverse effects in subjects in the treatment arm versus placebo at week 1-12 | Up to 12 weeks
Change from baseline at week 12 on the Columbia-Suicide Severity Rating Scale (C-SSRS) | baseline and at 12 weeks
Change from baseline at week 12 on the Arizona Sexual Experience (ASEX) scale | baseline and at 12 weeks

OTHER OUTCOMES:
Reduction of anxiety symptoms at 12 weeks as assessed by the Generalized Anxiety Disorder-7-item (GAD-) | at 12
Reduction of post traumatic stress symptoms at 12 weeks as assessed by the Post traumatic stress disorder Checklist for DSM-5 (PCL-5) | at 12 weeks
Improvement in sleep symptoms at 12 weeks as assessed by the Pittsburgh Sleep Quality Index (PSQI) | at 12 weeks
Reduction of aggressive symptoms at 12 weeks as assessed by the Modified Overt Aggression Scale (MOAS) | at 12 weeks
Improvement in cognition at 12 weeks as assessed by a composite z-score of the Rey Auditory Verbal Learning Test (RAVLT) score | at 12 weeks
Improvement in behavioral symptoms at 12 weeks as assessed by the Neuropsychiatric Inventory-Questionnaire (NPI-Q | at 12 weeks
Improvement in cognition at 12 weeks as assessed by a composite z-score of the Digit symbol substitution test (DSST) score | at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vani Rao, MD, Principal Investigator — Johns University and School of Medicine

IPD SHARING:
Plan to Share IPD: No
Prior to the initiation of the study, a method will be developed for data collection. Each participant will have a study folder with a unique identifying number to contain the results of study tests and evaluations. Another folder will also be kept that will hold all consent forms and identifying demographic information. The folders will be reviewed monthly for inconsistencies. The data will be entered into a database maintained in the Neuropsychiatry Division of Johns Hopkins Bayview Medical Center, which is password protected and only the PI and her Research team will have access to the study folders and database.
  The data monitoring committee will include Dr. Rao (PI), and members of the Data & Safety monitoring board: Drs. Christopher Marano, Paul Rosenberg and Jin Joo. All members of the Diagnostic and Statistical Manual of Mental Disorders (DSM) board are psychiatrists and faculty Johns Hopkins University. The 3 DSM members are not connected with the study.